CLINICAL TRIAL: NCT03266705
Title: A Phase 1, Open-label, Randomized, Crossover, Multiple Dose, Pivotal Bioequivalence Study To Compare Pf-06291826 4 X 20 Mg Tafamidis Meglumine And 61 Mga Tafamidis Free Acid Soft Gelatin Capsules Administered Under Fasted Conditions To Healthy Volunteers
Brief Title: A Study Comparing Amounts of 2 Different Forms of Tafamidis (PF-6291826) in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3461056; 2017-002572-15 (EudraCT Number)
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Healthy
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 61 mgA tafamidis free acid soft gelatin capsule (Experimental)
  Interventions: Drug: tafamidis
- 4x20 mg tafamidis meglumine soft gelatin capsule (Experimental)
  Interventions: Drug: tafamidis

INTERVENTIONS:
Drug: tafamidis — bioequivalence study

SUMMARY:
2 different formulations and doses of tafamidis will be compared. All subjects will receive both doses/formulations. Subjects will take tafamidis for 7 days, on the first 2 days they will take tafamidis twice, 12 hours apart and then once a day for the next 5 days. Subjects will be fasted before taking the drug. Blood samples will be taken to measure the amount of tafamidis starting on day 7 and ending on day 8. At least 16 days after the first formulation/dose is given, all subjects will repeat the procedure with the other formulation/dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males of females of non-childbearing potential
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* Blood pressure at screening visit of greater than 140 mm Hg (systolic) or 90 mg Hg (diastolic).
* Use of prescription or nonprescription drugs supplements within 7 days prior to 7 days of the study.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer)
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) | 24 hours
maximum observed plasma concentration (Cmax) | 24 hours

SECONDARY OUTCOMES:
minimum observed plasma concentration (Cmin) | 24 hours
Time to maximum observed plasma concentration (Tmax) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3461056&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Crossover%2C+Multiple+Dose%2C+Pivotal+Bioequivalence+Study+To+Compare+Pf-06291826+4+X+20+Mg+Tafamidis+Meglumine+And+61+Mga+Tafamidis+Free+Acid+Soft+Gelatin+Capsules+Administered+Under+Fasted+Conditions+To+Healthy+Volunteers